CLINICAL TRIAL: NCT02190526
Title: Therapeutic Effects of Mesalamine and Amitriptyline in IBS: a Randomized Clinical Trial
Brief Title: Effects of Mesalamine and Amitriptyline on Irritable Bowel Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study stopped due to lack of volunteer patients.
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8811215278
Record Dates: First submitted 2014-03-27; First posted 2014-07-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Diarrhea- Predominant Irritable Bowel Syndrome; Quality of Life
Keywords: mesalamine; amitriptyline; Severity of Illness Index
MeSH Terms: interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mesalazine(asacol 800 mg) (Experimental): patients receive asacol (800 mg/TDS) and a placebo agent similar to amitriptyline (10 mg/HS) for 8 weeks
  Interventions: Drug: Mesalazine(asacol 800 mg); Drug: placebo like amitriptyline
- Amitriptyline (Experimental): patients receive amitriptyline (10 mg/HS) and a placebo like asacol (800 mg/ TDS) for 8 weeks
  Interventions: Drug: Amitriptyline; Drug: placebo like asacol
- placebo group (Placebo Comparator): patients receive placebo like asacol (800 mg/TDS) and placebo similar to amitriptyline (10 mg/HS) for 8 weeks
  Interventions: Drug: placebo like asacol; Drug: placebo like amitriptyline

INTERVENTIONS:
Drug: Mesalazine(asacol 800 mg)
  Arms: Mesalazine(asacol 800 mg)
Drug: Amitriptyline
  Arms: Amitriptyline
Drug: placebo like asacol
  Arms: Amitriptyline; placebo group
Drug: placebo like amitriptyline
  Arms: Mesalazine(asacol 800 mg); placebo group

SUMMARY:
The aim of this study is to evaluate the effects of Mesalamine and Amitriptyline drugs on the Quality of Life and Symptom Severity Scale in patients with Diarrhea- Predominant Irritable Bowel Syndrome (IBS-D).

All patients will fill three validated questionnaires (IBS Symptom Severity Scale (IBS-SSS) , Hospital Anxiety and Depression Scale (HADS ) and IBS Quality of Life (IBS-QOL) ) at the beginning of trial and at weeks 2,4,6 and 8 of treatment.

Serum Immune Bio markers will be measured at 0,4, and 8 weeks of treatment. This study is a clinical trial upon 90 patients with Diarrhea- Predominant IBS (IBS-D) who are referred for the first time to our private gastrointestinal clinic from 2014 until 2016.

All patients who meet the inclusion criteria enrolled for a 2-week period screening phase. In order to exclude patients with Lactose intolerance, all patients take a lactose-free diet for 14 days before inclusion and patients whose symptoms improve by this regimen will be excluded.

This trial is a double-blind study and all patients will be assigned randomly to three groups:

1. Mesalazine group: Patients receive Asacol (800 mg/TDS) and a placebo agent similar to Amitriptyline (10 mg/HS) for 8 weeks
2. Amitriptyline group: Patients receive Amitriptyline (10 mg/HS) and a placebo like Asacol (800 mg/ TDS) for 8 weeks
3. Control group (placebo group): Patients receive placebo like Asacol (800 mg/TDS) and placebo similar to Amitriptyline (10 mg/HS) for 8 weeks

Ethical considerations:

1. All patients will fulfill an informed consent
2. Drugs are available without any charge
3. Observation of Helsinki ethical statement

ELIGIBILITY:
Inclusion Criteria:

1. Establishment of diagnosis of IBS by ROME-III criteria
2. Age > 18 years old and < 65 years old
3. Normal colonoscopy or sigmoidoscopy
4. Negative celiac serologic markers
5. Normal complete blood count (CBC) and stool exam and stool culture
6. The patient should not be administered Anti-inflammatory drugs such as Nonsteroidal Antiinflammatory Drugs(NSAIDs), oral or parenteral Antibiotics, Corticosteroids, Mast cell stabilizers, Narcotics, Antidepressants and Immunosuppressive Agents.
7. Normal thyroid-stimulating hormone (TSH )
8. Normal Serum Calcium
9. Educated patient

Exclusion Criteria:

1. Breast feeding and Pregnancy
2. Presence of acute or chronic inflammation which can change the basal level of cytokines
3. Allergic disorders like Asthma (family and personal history)
4. Presence of organic disease like Diabetes mellitus or Psychiatric disorders.
5. Alcohol dependency and addiction to Tobacco and Opium
6. Patients who do not use efficient contraception method
7. History of extensive abdominopelvic surgery except Appendectomy, Cholecystectomy, Hysterectomy and Cesarian-Section
8. Presence of Celiac disease
9. History of Crohn's disease, Ulcerative Colitis and Diverticulitis during the previous year.
10. History of Cardiac, Pulmonary, Hepatic and Renal disease
11. Presence of chronic GI disorders
12. History of Allergy to Aspirin, Mesalamine or Sulpha compounds
13. History of Lymphocytic or Microscopic Colitis
14. History of significant weight loss ( 10% of body weight during 6 months), nocturnal sweating, GI bleeding and family history of Colon cancer
15. Patients with Lactose intolerance disease
16. Presence of Bowel Acid Malabsorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
quality of life | 1 year
  All patients will fill three validated questionnaires (IBS-SSS , HADS and IBS-QOL ) at the beginning of trial and at weeks 2,4,6 and 8 of treatment to assess quality of life and symptom severity scale in patients with diarrhea- predominant .

SECONDARY OUTCOMES:
Serum immune biomarkers | 1 year
  Serum immune biomarkers will be measured at 0,4, and 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Ebrahimi Daryani, Professor, Study Director — Tehran University of Medical Science; Zahra Azizi, Researcher, Principal Investigator — Iran University of Medical Sciences; Mohammad Bashashati, Research Associate, Study Director — University of Calgary; Nima Rezaei, Assistant Professor, Study Director — Tehran University Of Medical Science
Locations (1):
- Gastrointestinal Private Clinic, Tehran, Tehran Province, Iran